CLINICAL TRIAL: NCT00973687
Title: Dexamethasone Tolerability in the Treatment of Acute Asthma in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: IWK Foundation (Unknown)
Responsible Party: Dr. Lyn Sonnenberg, IWK Health Centre
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2967
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2009-09

CONDITIONS: Asthma
Keywords: pediatric; dexamethasone; management; corticosteroids; asthma
MeSH Terms: conditions — Asthma | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 10 mg/mL Unsweetened Formulation (Placebo Comparator): no prior vomiting
  Interventions: Drug: Dexamethasone
- 1 mg/mL Ora Sweet Formulation (Experimental): no prior vomiting
  Interventions: Drug: Ora Sweet; Drug: Dexamethasone
- 10 mg/mL Unsweetened with prior vomiting (Active Comparator): with prior vomiting
  Interventions: Drug: Dexamethasone
- 1 mg/mL Ora Sweet with prior vomiting (Experimental): with prior vomiting
  Interventions: Drug: Ora Sweet; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ora Sweet — A pharmaceutical suspending vehicle and flavouring agent added to the dexamethasone. All arms received the same amount of dexamethasone based on the child's weight, only in different volumes.
  Arms: 1 mg/mL Ora Sweet Formulation; 1 mg/mL Ora Sweet with prior vomiting
Drug: Dexamethasone

SUMMARY:
The purpose of this study is to assess whether smaller volumes of oral dexamethasone result in better tolerability, specifically less vomiting, in pediatric patients during an acute asthma exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* acute asthma exacerbation
* requiring oral systemic corticosteroids for management

Exclusion Criteria:

* preference for pills over liquid formulation
* history of Nissen fundoplication surgery
* needed immediate airway intervention
* require oral medications to be given via a G or J tube
* if patient care would be compromised
* enrolled in the study on a previous visit.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 430 (Actual)
Dates: Start 2004-09; Primary Completion 2006-04 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study was to assess whether smaller volumes of oral dexamethasone resulted in better tolerability, specifically less vomiting, in pediatric patients with an acute exacerbation of asthma. | During Emergency Department visit

SECONDARY OUTCOMES:
To evaluate asthma symptom control post emergency room visit for acute asthma exacerbation. | 7-14 days following emergency dept visit

CONTACTS AND LOCATIONS:
Overall Officials: Lyn K Sonnenberg, MD, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada